CLINICAL TRIAL: NCT07215130
Title: Selective Removal of Endometriotic Lesions Using CUSA Clarity in Ovarian Endometriomas: A Case-Based Histopathological Study
Brief Title: Selective Removal of Endometriotic Lesions Using CUSA Clarity in Ovarian Endometriomas
Acronym: CUSA-ENDO
Status: Recruiting | Type: Observational
Sponsor: Kanazawa University (Other)
Responsible Party: Principal Investigator, Takashi IIZUKA, Doctor, Kanazawa University
Other Study IDs: KU-OBGYN-CUSA-2025-01
Record Dates: First submitted 2025-10-01; First posted 2025-10-10 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Ovarian Endometrioma; Endometriosis
Keywords: Endometriosis; Ovarian Cyst; CUSA Clarity; Ultrasonic Surgical Aspirator; Fertility Preservation; Histopathology
MeSH Terms: conditions — Endometriosis; Ovarian Cysts

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Formalin-fixed, paraffin-embedded (FFPE) tissue specimens of ovarian endometrioma cyst walls obtained during surgery. Samples will be used for histopathological and immunohistochemical analyses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ovarian Endometrioma Cases: Patients with ovarian endometriomas undergoing surgical excision at Kanazawa University Hospital. Cyst wall specimens are collected and analyzed ex vivo using the Cavitron Ultrasonic Surgical Aspirator (CUSA) Clarity device at different Tissue Select settings. Histopathological evaluation is performed to assess selective removal of endometriotic epithelium and preservation of ovarian stroma.
  Interventions: Device: Cavitron Ultrasonic Surgical Aspirator (CUSA) Clarity

INTERVENTIONS:
Device: Cavitron Ultrasonic Surgical Aspirator (CUSA) Clarity — Ex vivo application of the Cavitron Ultrasonic Surgical Aspirator (CUSA) Clarity device to ovarian endometrioma cyst wall specimens. Tissue Select settings from 0 to 4 are used to evaluate tissue selectivity, specifically removal of endometriotic epithelium while preserving normal ovarian stroma. Samples are subsequently analyzed histopathologically.
  Other Names: CUSA Clarity

SUMMARY:
This study aims to evaluate the feasibility and tissue selectivity of a novel surgical technology, the Cavitron Ultrasonic Surgical Aspirator (CUSA) Clarity, in the management of ovarian endometriomas. Ovarian endometriomas are cysts caused by endometriosis that can damage ovarian reserve when treated by conventional surgery. In this study, ovarian cyst wall specimens are examined ex vivo using different Tissue Select settings of the CUSA device. Histopathological analyses are performed to determine whether endometriotic epithelium can be selectively removed while preserving normal ovarian tissue. The findings may contribute to developing fertility-preserving surgical approaches for women with endometriomas.

DETAILED DESCRIPTION:
Endometriomas are one of the most common manifestations of endometriosis and are frequently associated with infertility. Conventional cystectomy often results in inadvertent removal of normal ovarian tissue, which may reduce ovarian reserve. To address this issue, the Cavitron Ultrasonic Surgical Aspirator (CUSA) Clarity system, particularly with the Tissue Select mode, has been proposed as a tissue-selective surgical device.

In this observational histopathological study, ovarian endometrioma wall specimens obtained during surgery are divided into multiple parts. Each part is subjected to ex vivo treatment with the CUSA Clarity device at different Tissue Select settings (0-4). The treated samples are fixed, paraffin-embedded, and stained with hematoxylin-eosin and immunohistochemical markers (e.g., cytokeratin 7, CD10). Pathologists evaluate the extent of removal of endometriotic lesions and preservation of normal ovarian stroma.

The primary objective is to assess whether endometriotic epithelium can be selectively removed while sparing ovarian stromal tissue. Secondary objectives include evaluation of the depth of tissue removal and the presence of residual lesions at unscraped margins. The results are expected to provide histopathological evidence supporting the potential clinical application of CUSA in fertility-preserving surgery for ovarian endometriomas.

ELIGIBILITY:
Inclusion Criteria:

* Female patients diagnosed with ovarian endometrioma who undergo surgical treatment (cystectomy or adnexectomy) at Kanazawa University Hospital between January 1, 2025, and March 31, 2027.
* Written informed consent obtained prior to study participation.
* Age ≥ 20 years at the time of consent.
* For patients with previously stored endometrioma specimens under a broad consent, additional written consent for participation in this study will be obtained.

Exclusion Criteria:

* Patients with suspected malignancy based on preoperative imaging.
* Patients judged by the attending physician to be unsuitable for participation in this study for any reason.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women aged 20 years or older diagnosed with ovarian endometrioma and treated surgically at Kanazawa University Hospital. Surgically resected ovarian endometrioma specimens are used for ex vivo histopathological evaluation of selective lesion removal using the CUSA® Clarity device.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2025-01-30 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Histopathological confirmation of selective removal of endometriotic epithelium with preservation of ovarian stroma | Immediately after ex vivo CUSA treatment of specimens (within 1 day of surgery)
  Evaluation of hematoxylin-eosin and immunohistochemical stained sections to determine whether endometriotic epithelial lining is removed while normal ovarian stroma is preserved.

SECONDARY OUTCOMES:
Depth of tissue removal at different Tissue Select settings | Immediately after ex vivo treatment
  Histological measurement of tissue removal depth under Tissue Select settings 0-4 using H&E and Sirius Red staining.
Presence of residual endometriotic lesions at unscraped margins | Immediately after ex vivo treatment
  Histological evaluation of cyst wall margins not subjected to CUSA scraping to confirm lesion selectivity.
Immunohistochemical assessment of epithelial and stromal markers | Within 1 week after sample fixation and processing
  Immunostaining with cytokeratin 7 (epithelial) and CD10 (stromal) to assess selective tissue removal.

CONTACTS AND LOCATIONS:
Overall Officials: Kaoru Abiko, MD, PhD, Principal Investigator — Kanazawa University, Department of Obstetrics and Gynecology
Locations (1):
- Kanazawa University Hospital, Kanazawa, Ishikawa-ken, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Muzii L, Bianchi A, Bellati F, Cristi E, Pernice M, Zullo MA, Angioli R, Panici PB. Histologic analysis of endometriomas: what the surgeon needs to know. Fertil Steril. 2007 Feb;87(2):362-6. doi: 10.1016/j.fertnstert.2006.06.055. Epub 2006 Nov 13. PMID 17094980
- [Background] D'Alterio MN, Nappi L, Vitale SG, Agus M, Fanni D, Malzoni M, Falcone F, Sorrentino F, D'Agate MG, Scibilia G, Mereu L, Scollo P, Angioni S. Evaluation of Ovarian Reserve and Recurrence Rate After DWLS Diode Laser Ovarian Endometrioma Vaporization (OMAlaser): A Prospective, Single-Arm, Multicenter, Clinical Trial. J Minim Invasive Gynecol. 2025 Mar;32(3):279-287. doi: 10.1016/j.jmig.2024.10.021. Epub 2024 Oct 28. PMID 39477011
- [Background] Ferrari SM, Dolci C, Taccagni G, Congia C, Ottolina J, Schimberni M, Bartiromo L, Candiani M. Histologic findings from ablation of ovarian endometriomas using argon plasma coagulation (APC-ENDO): a pilot study. Eur J Obstet Gynecol Reprod Biol. 2025 Aug;312:114532. doi: 10.1016/j.ejogrb.2025.114532. Epub 2025 Jun 14. PMID 40540997
- [Background] Candiani M, Ottolina J, Posadzka E, Ferrari S, Castellano LM, Tandoi I, Pagliardini L, Nocun A, Jach R. Assessment of ovarian reserve after cystectomy versus 'one-step' laser vaporization in the treatment of ovarian endometrioma: a small randomized clinical trial. Hum Reprod. 2018 Dec 1;33(12):2205-2211. doi: 10.1093/humrep/dey305. PMID 30299482
- [Background] Younis JS, Shapso N, Ben-Sira Y, Nelson SM, Izhaki I. Endometrioma surgery-a systematic review and meta-analysis of the effect on antral follicle count and anti-Mullerian hormone. Am J Obstet Gynecol. 2022 Jan;226(1):33-51.e7. doi: 10.1016/j.ajog.2021.06.102. Epub 2021 Jul 13. PMID 34265271
- [Background] Muzii L, Di Tucci C, Di Feliciantonio M, Marchetti C, Perniola G, Panici PB. The effect of surgery for endometrioma on ovarian reserve evaluated by antral follicle count: a systematic review and meta-analysis. Hum Reprod. 2014 Oct 10;29(10):2190-8. doi: 10.1093/humrep/deu199. Epub 2014 Aug 1. PMID 25085800
- [Background] Vasquez JM, Eisenberg E, Osteen KG, Hickerson D, Diamond MP. Laparoscopic ablation of endometriosis using the cavitational ultrasonic surgical aspirator. J Am Assoc Gynecol Laparosc. 1993 Nov;1(1):36-42. doi: 10.1016/s1074-3804(05)80756-x. PMID 9050458
- [Background] Adamyan L, Kasyan V, Pivazyan L, Isaeva S, Avetisyan J. Laser vaporization compared with other surgical techniques in women with ovarian endometrioma: a systematic review and meta-analysis. Arch Gynecol Obstet. 2023 Aug;308(2):413-425. doi: 10.1007/s00404-022-06799-4. Epub 2022 Sep 29. PMID 36175684
- [Background] Matsuzaki S, Houlle C, Darcha C, Pouly JL, Mage G, Canis M. Analysis of risk factors for the removal of normal ovarian tissue during laparoscopic cystectomy for ovarian endometriosis. Hum Reprod. 2009 Jun;24(6):1402-6. doi: 10.1093/humrep/dep043. Epub 2009 Feb 26. PMID 19246468
- [Background] Bafort C, Beebeejaun Y, Tomassetti C, Bosteels J, Duffy JM. Laparoscopic surgery for endometriosis. Cochrane Database Syst Rev. 2020 Oct 23;10(10):CD011031. doi: 10.1002/14651858.CD011031.pub3. PMID 33095458
- See also: Official website of the Department of Obstetrics and Gynecology, Kanazawa University — https://kanazawa-obgyn.org/obgyn/index.html